CLINICAL TRIAL: NCT04843917
Title: Immunity Against the COVID-19 Vaccine in Healthcare Workers of Buenos Aires, Argentine.
Brief Title: Immunity Against COVID-19 Vaccine in Healthcare Workers in Argentine
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, VANINA LAURA PAGOTTO, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 3913
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Coronavirus 2019; Healthcare Workers; Vaccine
Keywords: COVID-19 Vaccines; Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immunoglobulin G detection — Detection of immunoglobulin G against Spike Receptor Binding Domain against severe acute respiratory syndrome coronavirus 2

SUMMARY:
Vaccination against coronavirus disease 19 (COVID-19) is an essential primary prevention tool to limit the health and economic effects of the pandemic. Objectives: To determine the variation in the levels of Immunoglobulin G (IgG) antibodies in health workers who received a COVID-19 vaccine.

DETAILED DESCRIPTION:
Vaccination against coronavirus disease 19 (COVID-19) is an essential primary prevention tool to limit the health and economic effects of the pandemic. The Ministry of Health of the Nation, designed the "Strategic Plan for vaccination", which the first line being the health workers " The National Administration of Medicines, Food and Medical Technology authorized two emergency vaccines for administration, Sputnik V and Sinopharm vaccine. It is important to evaluate immunogenicity and its correlation with the long-term efficacy and safety profile of this vaccines.

Objectives: To determine the variation in the levels of Immunoglobulin G (IgG) antibodies in health workers who received a COVID-19 vaccine between the time before the first dose, and after 1 month, 6 months and 12 months after the completion of the immunization, depending on whether they have received the Sputnik V vaccine or the Sinopharm vaccine, and correlate the Immunoglobulin G levels with the presence of adverse events and infection with COVID-19 Methodology: Design: observational and analytical study of a prospective cohort of healthcare workers immunized with some COVID-19 vaccine. The presence of IgG will be determined qualitatively and quantitatively. The immunoglobulin G titer in each period will be compared globally and according to the type of vaccine administered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects receiving any COVID-19 vaccine.

Exclusion Criteria:

* Subjects who do not agree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers who want to receive any COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
To assess the change in the levels of Immunoglobulin G (IgG) antibodies from baseline at 1 month, at 6 months and at 12 months after the completion of the immunization in health workers who received a COVID-19 vaccine | 1 year
  To assess the change in the levels of Immunoglobulin G (IgG) antibodies from baseline at 1 month, at 6 months and at 12 months after the completion of the immunization in health workers who received a COVID-19 vaccine
To correlate the Immunoglobulin G levels with the presence of adverse events and infection with COVID-19 | 1 year
  To correlate the Immunoglobulin G levels with the presence of adverse events and infection with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: vanina Pagotto, MSC, Principal Investigator — Hospital Italiano de Buenos Aires; Silvana Figar, MSC, Study Chair — Hospital Italiano de Buenos Aires; Hernán Garcia Rivello, Pharm, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Logunov DY, Dolzhikova IV, Zubkova OV, Tukhvatullin AI, Shcheblyakov DV, Dzharullaeva AS, Grousova DM, Erokhova AS, Kovyrshina AV, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Lubenets NL, Egorova DA, Shmarov MM, Nikitenko NA, Morozova LF, Smolyarchuk EA, Kryukov EV, Babira VF, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine in two formulations: two open, non-randomised phase 1/2 studies from Russia. Lancet. 2020 Sep 26;396(10255):887-897. doi: 10.1016/S0140-6736(20)31866-3. Epub 2020 Sep 4. PMID 32896291
- [Result] Logunov DY, Dolzhikova IV, Shcheblyakov DV, Tukhvatulin AI, Zubkova OV, Dzharullaeva AS, Kovyrshina AV, Lubenets NL, Grousova DM, Erokhova AS, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Egorova DA, Shmarov MM, Nikitenko NA, Gushchin VA, Smolyarchuk EA, Zyryanov SK, Borisevich SV, Naroditsky BS, Gintsburg AL; Gam-COVID-Vac Vaccine Trial Group. Safety and efficacy of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine: an interim analysis of a randomised controlled phase 3 trial in Russia. Lancet. 2021 Feb 20;397(10275):671-681. doi: 10.1016/S0140-6736(21)00234-8. Epub 2021 Feb 2. PMID 33545094
- [Result] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Result] Di Pasquale A, Bonanni P, Garcon N, Stanberry LR, El-Hodhod M, Tavares Da Silva F. Vaccine safety evaluation: Practical aspects in assessing benefits and risks. Vaccine. 2016 Dec 20;34(52):6672-6680. doi: 10.1016/j.vaccine.2016.10.039. Epub 2016 Nov 8. PMID 27836435
- [Result] Herve C, Laupeze B, Del Giudice G, Didierlaurent AM, Tavares Da Silva F. The how's and what's of vaccine reactogenicity. NPJ Vaccines. 2019 Sep 24;4:39. doi: 10.1038/s41541-019-0132-6. eCollection 2019. PMID 31583123
- [Result] Virtanen M, Peltola H, Paunio M, Heinonen OP. Day-to-day reactogenicity and the healthy vaccinee effect of measles-mumps-rubella vaccination. Pediatrics. 2000 Nov;106(5):E62. doi: 10.1542/peds.106.5.e62. PMID 11061799
- [Result] Mitchell TC, Casella CR. No pain no gain? Adjuvant effects of alum and monophosphoryl lipid A in pertussis and HPV vaccines. Curr Opin Immunol. 2017 Aug;47:17-25. doi: 10.1016/j.coi.2017.06.009. Epub 2017 Jul 17. PMID 28728074
- [Result] Sadoff J, Le Gars M, Shukarev G, Heerwegh D, Truyers C, de Groot AM, Stoop J, Tete S, Van Damme W, Leroux-Roels I, Berghmans PJ, Kimmel M, Van Damme P, de Hoon J, Smith W, Stephenson KE, De Rosa SC, Cohen KW, McElrath MJ, Cormier E, Scheper G, Barouch DH, Hendriks J, Struyf F, Douoguih M, Van Hoof J, Schuitemaker H. Interim Results of a Phase 1-2a Trial of Ad26.COV2.S Covid-19 Vaccine. N Engl J Med. 2021 May 13;384(19):1824-1835. doi: 10.1056/NEJMoa2034201. Epub 2021 Jan 13. PMID 33440088
- [Result] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Result] Hope JL, Bradley LM. Lessons in antiviral immunity. Science. 2021 Jan 29;371(6528):464-465. doi: 10.1126/science.abf6446. No abstract available. PMID 33510014
- See also: World Health Organization. COVID-19 vaccines — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/covid-19-vaccines
- See also: National Drug, Food, and Medical Technology Administration report on the Sputnik V vaccine — https://www.argentina.gob.ar/noticias/informe-de-la-anmat-sobre-la-vacuna-sputnik-v
- See also: Ministry of Health, Argentina. COVID-19 vaccine — https://www.argentina.gob.ar/coronavirus/vacuna
- See also: Ministry of Health, Argentina. Strategic Plan for vaccination against COVID-19 in Argentina — https://www.argentina.gob.ar/coronavirus/vacuna/plan-estrategico
- See also: Active surveillance of the sputnik v vaccine in health workers — https://doi.org/10.1101/2021.02.03.21251071
- See also: Bank of Communication Resources of the Ministry of Health of the Nation. Fifth Vaccine Safety Report — https://bancos.salud.gob.ar/recurso/quinto-informe-de-seguridad-en-vacunas